CLINICAL TRIAL: NCT00797719
Title: A Feasibility Study Evaluating Neoadjuvant Hemithoracic Intensity Modulated Radiation Therapy for Surgically Resectable Malignant Pleural Mesothelioma
Brief Title: Short Neoadjuvant Hemithoracic IMRT for MPM
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 08-0106-C
Record Dates: First submitted 2008-11-21; First posted 2008-11-25 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: MPM; Short hemithoracic IMRT
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All (Experimental): This is a single arm study. All patients enrolled will be in this arm.
  Interventions: Other: Pre-op RT +/- chemotherapy

INTERVENTIONS:
Other: Pre-op RT +/- chemotherapy — Patients on the study will receive IMRT for approximately 1 week of 5 daily treatments. Short pre-operative hemithoracic RT is a new technique. 1 week post-RT, they will proceed with an extrapleural pneumonectomy. If the mediastinal lymph nodes that are removed during surgery are positive for tumour cells, 3 cycles of chemotherapy, consisting of raltitrexed and cisplatin, will be given 6-12 weeks post-surgery.

SUMMARY:
Malignant pleural mesotheliomas (MPMs) are tumours associated with asbestos exposure involving the tissue lining surrounding the lung. Radiation therapy (RT) dramatically reduces the risk of tumour recurrence within the irradiated area (>90%). But patients continue to succumb to MPMs due to the tumour spreading outside the chest cavity. This may be due to tumour cells inadvertently contaminating areas outside the chest cavity during surgery. The study will look at whether giving a short intense course of chest radiation just prior to surgery will sterilized these tumour cells and thus, avoid or reduce contamination of the areas outside the chest cavity. The investigators hypothesize that short neoadjuvant (pre-operative) hemithoracic RT, followed by immediate planned extrapleural pneumonectomy (EPP) (+/- adjuvant chemotherapy) will reduce the risk of intra-operative seeding and reduce the incidence of distant metastatic disease.

DETAILED DESCRIPTION:
The study is a phase I/II prospective single cohort clinical feasibility study. 100 patients with early stage resectable malignant pleural mesothelioma will be enrolled into the study. Patients will have a baseline PET scan. Patients on the study will receive IMRT for approximately 1 week of 5 daily treatments. 1 week post-RT, they will proceed with an extrapleural pneumonectomy. If the mediastinal lymph nodes that are removed during surgery are positive for tumour cells, 3 cycles of chemotherapy, consisting of raltitrexed and cisplatin OR Pemetrexed and cisplatin, will be given 6-12 weeks post-surgery. Before and during treatment, side effects will be assessed. After treatment, follow up visits will be conducted every 1 to 2 months for the first year, and every 3 months for the second year. At each visit, a history and physical examination will be performed and ECOG performance status will be assessed. Routine tests will include CBC, liver profile, creatinine and chest x-ray. CT thorax and abdomen will be done at 3, 6, 12, 18, and 24 months. Additional test may be done at the discretion of the oncologist if the patient becomes symptomatic. The study will evaluate the feasibility and safety of short pre-operative RT, and may help confirm the intraoperative seeding hypothesis. Preoperative RT may also reduce the risk of both local and distant spread and, ultimately, improve overall survival. By shortening overall treatment time, it may also improve patient compliance and convenience. We may be able to give chemotherapy only to patients that are at highest risk and avoid it in others.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status of 0-2
* Good pulmonary function precluding radiation therapy (FEV>1 L or >40% predicted or DLCO >45% predicted)
* Any patient wiht a new histological diagnosis of malignancy pleural mesothelioma (MPM). Sarcomatoid or biphasic histologies can be included but will be analyzed separately due to their poor prognosis
* Stage T1-2N0M0 based on conventional investigations and tests. Selected stage T3N0M0 may be included at the discretion of the surgeon if deemed resectable.
* Suitable for combined modality therapy
* Informed consent

Exclusion Criteria:

* Distant metastatic disease
* Previous thoracic irradiation
* Serious non-malignant disease (e.g. cardiovascular, pulmonary, systemic lupus erythematosus (SLE), scleroderma) which would preclude definitive radiation treatment
* Previous chemotherapy for this or concurrent malignancy
* Previous concomitant malignancies except for patients with non-melanoma skin cancer, contralateral non-invasive breast cancer, prostate cancer treated with curative intent or carcinoma in situ of any other site. In addition, patients with invasive cancers treated more than 3 years previously and without evidence of recurrence will be eligible
* Women who are currently pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-10 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome for the study will be the proportion of patients treated as per protocol without treatment related mortality. | After completion of therapy: every 4 wks for 3 mos, then every 6 wks for 6 mos, then every 2 mos for 12 mos, then every 3 mos for 2 yrs, then every 6 mos for 5 years

SECONDARY OUTCOMES:
To evaluate: acute and late morbidity related to treatment; local & distant recurrence, disease free & overall survival; identify factors/parameters associated with increased risk of treatment morbidity | After completion of therapy: every 4 wks for 3 mos, then every 6 wks for 6 mos, then every 2 mos for 12 mos, then every 3 mos for 2 yrs, then every 6 mos for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Cho, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Chan M, Wu L, Yun Z, McKee TD, Cabanero M, Zhao Y, Kohno M, Murakami J, de Perrot M. Blocking the GITR-GITRL pathway to overcome resistance to therapy in sarcomatoid malignant pleural mesothelioma. Commun Biol. 2021 Jul 26;4(1):914. doi: 10.1038/s42003-021-02430-5. PMID 34312483
- [Derived] Cho BCJ, Donahoe L, Bradbury PA, Leighl N, Keshavjee S, Hope A, Pal P, Cabanero M, Czarnecka K, McRae K, Tsao MS, de Perrot M. Surgery for malignant pleural mesothelioma after radiotherapy (SMART): final results from a single-centre, phase 2 trial. Lancet Oncol. 2021 Feb;22(2):190-197. doi: 10.1016/S1470-2045(20)30606-9. Epub 2021 Jan 12. PMID 33450184
- [Derived] de Perrot M, Dong Z, Bradbury P, Patsios D, Keshavjee S, Leighl NB, Hope A, Feld R, Cho J. Impact of tumour thickness on survival after radical radiation and surgery in malignant pleural mesothelioma. Eur Respir J. 2017 Mar 15;49(3):1601428. doi: 10.1183/13993003.01428-2016. Print 2017 Mar. PMID 28298401
- [Derived] Cho BC, Feld R, Leighl N, Opitz I, Anraku M, Tsao MS, Hwang DM, Hope A, de Perrot M. A feasibility study evaluating Surgery for Mesothelioma After Radiation Therapy: the "SMART" approach for resectable malignant pleural mesothelioma. J Thorac Oncol. 2014 Mar;9(3):397-402. doi: 10.1097/JTO.0000000000000078. PMID 24445595